CLINICAL TRIAL: NCT01549392
Title: Feasibility Study of Magnetic Resonance Spectroscopy and Dynamic Enhanced Cat Scan Imaging in Glioblastomas Treated With and Without Avastin
Brief Title: Imaging Study of Glioblastomas Treated With Avastin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient accrual
Sponsor: London Health Sciences Centre (Other)
Collaborators: University of Western Ontario, Canada (Other); London Regional Cancer Program, Canada (Other)
Responsible Party: Principal Investigator, Barbara Fisher, Dr, London Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LRCP02
Record Dates: First submitted 2012-02-17; First posted 2012-03-09 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Malignant Gliomas
Keywords: dynamic enhanced ct scan; mri spectroscopy; recurrent gliomas
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DECT/MR Spectroscopy +Avastin (Active Comparator): -15 Glioma Patients with progression will undergo DECT and MRS before Avastin (10 mg/kg iv q2 weeks until progression) and 3 months later
  Interventions: Device: DECT; Device: MR spectroscopy
- DECT/MR Spectroscopy no Avastin (Active Comparator): 15 glioma patients not receiving Avastin for recurrence studied in the same manner as Arm 1
  Interventions: Device: DECT; Device: MR spectroscopy

INTERVENTIONS:
Device: DECT — DECT at tumor progression and 3 months later
  Other Names: 3 T 64-slice CT scanner (Discovery CT750 HD, GE Healthcare
Device: MR spectroscopy — MR spectroscopy at tumor progression and 3 months later
  Other Names: MRI scanner: Siemens 3T Tim Trio; Sequences: T1W, DTI; Analysis software: Brain voyager

SUMMARY:
This study aims to assess the effect of Avastin on brain vascularity and blood-brain permeability using dynamic contrast ct scans (DECT) and MRI imaging. Previous publications have documented the method by which DECT can determine alterations in vascular volume and tissue permeability within tumors and normal brain tissue. Functional maps of cerebral blood flow cerebral blood volume and permeability-surface area can be generated from the DECT studies to assess tumor perfusion. MRI spectroscopy analyzes brain chemistry to detect tumour versus edema versus normal brain. Thirty patients will receive MRI spectroscopy and DECT imaging at the time of presumed recurrence and 3 months later. 15 patients who do not receive Avastin and 15 patients who do receive Avastin as standard treatment for recurrence will be studied with DECT and MRI spectroscopy at baseline and then again in 3 months.

DETAILED DESCRIPTION:
The clinical determination of the point of tumour progression or response is difficult to determine using standard diagnostic imaging ie CT/MRI especially following previous treatment with surgery, radiation and chemotherapy. Hemorrhage, edema, inflammation and vascular necrosis.

Both MR spectroscopy and DECT have been reported as being able to define areas of recurrent tumour as opposed to treatment-related effects. We wish to investigate the correlation between MR spectroscopy and DECT in assessing tumour progression or response to Avastin in comparison with patients not receiving Avastin.

Health Canada has approved Avastin for clinical use in patients with recurrent glioblastoma who have previously received temozolomide and radiotherapy. We propose to perform a DECT scan at baseline at presumed tumour progression and again 3 months to determine the effects of tumour progression/response on blood brain barrier permeability and vascular volume. The group of 15 patients will be compared to a group of 15 patients who do not receive Avastin at recurrence involving DECT scanning and MR spectroscopy at the time of the radiological progression and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of glioblastoma with clinical or radiological evidence of progression as indicated by the RANO criteria 19
* Previous radiation and temozolomide chemotherapy
* Patients must be receiving Avastin chemotherapy as second-line treatment if in the Avastin group
* Study-specific consent

Exclusion Criteria:

* Failure to meet inclusion criteria
* Pregnant or lactating patients
* Allergy to iodine or CT contrast precludes DECT component of study
* Claustrophobia precludes MR Spectroscopy component of study
* Internal metal which would preclude an MRI scan

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Fisher, MD, Principal Investigator — London Regional Cancer Program
Locations (1):
- London Regional Cancer Centre, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- DECT/MRS in Patients Receiving Avastin: 3 Glioma Patients underwent DECT and MRS pre-Avastin and 3 months later after receiving avastin 10 mg/kg iv q2weeks
  DECT: DECT at tumor progression and 3 months later
  MR spectroscopy: MR spectroscopy at tumor progression and 3 months later Avastin 10 mg/kg iv q2weeks
- DECT/MRS in Glioma Patients Not Receiving Avastin: 0 glioma patients not receiving Avastin for recurrence studied in the same manner as Arm 1
  DECT: DECT at tumor progression and 3 months later
  MR spectroscopy: MR spectroscopy at tumor progression and 3 months later
Period: Overall Study
Arm/Group | DECT/MRS in Patients Receiving Avastin | DECT/MRS in Glioma Patients Not Receiving Avastin
Started | 3 | 0
Completed | 2 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: patients with recurrent glioblastoma
Groups:
- DECT/MRS in Patients Receiving Avastin: -15 Glioma Patients with progression will undergo DECT and MRS pre-Avastin and 3 months later
  DECT: DECT at tumor progression and 3 months later
  MR spectroscopy: MR spectroscopy at tumor progression and 3 months later
- DECT/MRS in Glioma Patients Not Receiving Avastin: 15 glioma patients not receiving Avastin for recurrence studied in the same manner as Arm 1
  DECT: DECT at tumor progression and 3 months later
  MR spectroscopy: MR spectroscopy at tumor progression and 3 months later
- Total: Total of all reporting groups
Arm/Group | DECT/MRS in Patients Receiving Avastin | DECT/MRS in Glioma Patients Not Receiving Avastin | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 50 [45 to 65] |  | 50 [45 to 65]
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: 3 Month Response
Description: participants who had reduction of tumor size from avastin at 3 months
Time Frame: at 3 months after initial DECT and MR spectroscopy
Measure: Number; unit: participants who had tumor reduction
Arm/Group | DECT/MRS in Patients Receiving Avastin | DECT/MRS in Glioma Patients Not Receiving Avastin
Number analyzed (Participants) | 3 | 0
participants who had tumor reduction | 3 |

ADVERSE EVENTS:
Arm/Group | DECT/MRS in Patients Receiving Avastin | DECT/MRS in Glioma Patients Not Receiving Avastin
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No